CLINICAL TRIAL: NCT02443272
Title: A Randomized Comparison Study of Minimally Invasive Loop Drainage Versus Standard Incision and Drainage for Skin Abscesses in Children
Brief Title: Comparison of Loop Drainage Versus Incision and Drainage for Abscesses in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seton Healthcare Family (Other)
Collaborators: Scientific, Education and Research Foundation of UTSW Austin (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR-14-114
Record Dates: First submitted 2015-05-11; First posted 2015-05-13 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-04

CONDITIONS: Abscess of Skin and/or Subcutaneous Tissue
MeSH Terms: interventions — Drainage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Arm (Active Comparator): Receive standard incision and drainage
  Interventions: Procedure: Incision and Drainage
- Intervention Arm (Experimental): Receive minimal invasive loop drainage using the Vesi-loop device
  Interventions: Procedure: Vessel Loop Drainage

INTERVENTIONS:
Procedure: Vessel Loop Drainage — Minimally invasive approach will utilize a vesi-loop device for the vessel loop drainage technique by placing 2 peripheral stab incisions into the abscess with a tunnel through the abscess cavity, and loop passed through the tunnel and tied atop the skin.
  Arms: Intervention Arm
Procedure: Incision and Drainage — Standard of care treatment will utilize incision and drainage over the center of the abscess cavity with or without packing at physicians discretion.
  Arms: Control Arm

SUMMARY:
The purpose of this study is to compare abscess drainage utilizing the vessel loop technique in children to the standard incision and drainage technique with the endpoint to determine if rates of treatment failure are non-inferior.

DETAILED DESCRIPTION:
BACKGROUND INFORMATION:

Infections of skin and soft tissue remain one of the more common chief complaints in the pediatric emergency department. With methicillin-resistant Staphylococcus aureus being a prevalent pathogen, abscess development is not uncommon. The emergency department remains the common setting for required therapeutic intervention. However, active investigation exists in regard to the ideal intervention for children and adults.

Incision and drainage of cutaneous abscess has remained the standard of care for years. However this standard has been adopted without robust supportive evidence. Recently, various studies have questioned the benefit of various aspects of treatment, including antibiotics, incision size, and necessity for packing. Other studies have even suggested a less-invasive approach. Some of these have utilized a vessel loop and have demonstrated a reduced need for home-health visits, reduced inpatient length of stay, good patient tolerance, and no increase in failure rates. These studies are, however, retrospective in design with execution primarily by the surgical team.

STUDY DESCRIPTION:

Upon obtaining written informed consent/assent by the study team member, subjects will be randomized using a computerized randomization procedure and opaque envelopes. Initially, thorough history and physical exam will be performed. A data sheet will be completed detailing patient characteristics (eg. age, gender, ethnicity, prior treatment) and wound characteristics (eg. greatest diameter of both erythema and induration, presence of spontaneous drainage, location). Pain control/procedural sedation will be selected at the discretion of the treating physician, consistent with current local practice (eg. topical lidocaine, intranasal fentanyl and/or midazolam, oral acetaminophen/hydrocodone or ibuprofen, intravenous ketamine, morphine, or fentanyl). Pain will be assessed prior to physical exam and again shortly after the procedure via the validated FACES-Revised Pain Scale. The patient will provide this assessment if 5 years or older. Otherwise, the parent will provide the degree of pain perceived for their child. The difference between these two pain assessments will be evaluated as an endpoint. Physicians will report on their satisfaction with the procedure using a 5-point Likert scale.

The control arm of incision and drainage will require a single linear incision over the most fluctuant portion of the abscess at a length deemed necessary by the treating physician. Expressed contents will be sent for wound culture. Loculations will be disrupted with a hemostat followed by copious irrigation with sterile saline. At the discretion of the treating physician, the wound may be packed with ¼-inch iodoform gauze and dressed with dry gauze.

The intervention arm of vessel loop-drainage will require placement of a small incision of 4-5 mm at the periphery of induration. Expressed contents will be sent for wound culture. Using a hemostat, the loculations will be disrupted and expressed. Using the hemostat through the abscess cavity, the opposite aspect will be probed and a second 4-5 mm incision will be placed. The cavity will then be copiously irrigated with saline. A vessel loop (DeRoyal Industries; Powell, TN) will then be pulled through the cavity via the two incisions and loosely tied to itself above the skin using a surgeons knot. The wound will be dressed with dry gauze.

A prescription for antibiotics and pain medication will be provided at the discretion of the treating physician. The parent will be given standardized wound-care instructions (twice-daily soaks for 5 days with dry dressing re-application), contact information (phone and email) will be confirmed, selection of 24-48 hour follow-up will be made, and necessity of the 14- and 90-day follow-up will be emphasized. The parents will be encouraged to keep a pain medication diary (charted upon their care instructions) and bring the diary to their 2 initial follow-up appointments.

Upon completion of the initial ED encounter, data will be collected regarding type of pain control/procedural sedation during the ED course, selection of prescribed antibiotics and pain medication, and eventually results of wound culture.

24-48 hours after the incision and drainage procedure, subjects will return to the ED for a repeat evaluation. Packing will be removed from patients in the standard incision and drainage arm. The wound will be evaluated for five inflammatory components (i.e. presence of induration, fluctuance, drainage, tenderness, and warmth). If the evaluating physician decides that an abscess is still present and requires re-instrumentation, or if the infection requires admission for IV antibiotics, treatment failure will be declared. Following the assessment, the control arm may be repacked only if determined to be necessary. Parents will report on their satisfaction with the procedure, and simplicity of and anxiety with wound care utilizing a Likert scale of 1-5. Pain medication use will be quantified using their diary and then documented. Their contact information will be reconfirmed and the second follow-up appointment will be scheduled.

Subjects in the loop-drainage arm will receive emphasized instruction about technique and timing of loop removal. This will be performed at home only after drainage has ceased. Local practice by the general surgeon group suggests this is typically around post-operative day 5. Previous loop studies have performed this removal near day 8 to 10. We will encourage the parent to remove the loop on day 7 (if drainage has ceased) by simply cutting one side of the loop and pulling it from the cavity. A phone call will be performed on day 7 to assess readiness and provide support for removal. The day of loop removal will be documented.

Follow-up at post-procedure day 14 will be performed in the ED by a physician member of the study team. Prior to this visit, the parent will be reminded via telephone and email 2-3 days prior to the appointment. The wound will be evaluated for the same signs of inflammation as the previous visit. The wound will again be evaluated for indications of re-instrumentation or hospital admission (treatment failure). If the patient demonstrates systemic illness, parenteral antibiotics will be initiated with admission to the hospital. A second assessment will be performed at this follow-up visit; the Hollander scale will be applied to determine cosmetic outcome. The same Likert scales will be given to the parent regarding both the simplicity of, and anxiety with wound care. Pain medication use will again be quantified using their diary and then documented. The parent will be asked if any other physician encounters (here or elsewhere) were pursued and if re-instrumentation or hospital admission occurred. Follow-up will be encouraged with a $25 gift card (utilizing funding received from Scientific, Education and Research Foundation of UTSW Austin Research/Fellow Grant, and from research funds of the PEM fellowship department) to compensate families for their time and travel.

If the subject is unable to make the second follow-up appointment, a phone call will be performed to inquire if the patient presented to a hospital for intervention secondary to treatment failure of the initial abscess. If phone follow-up is unsuccessful, computerized chart review of the Seton network will be performed to obtain the same end-point.

At 3 months, parents will be called to inquire of their satisfaction with the wound scar using a 5-point Likert scale. They will also be reminded to return to the hospital to obtain photographic documentation of the scar. Another $25 gift card will be issued to those able to do so.

All patient records will be maintained in a locked, secure location, accessible by research personnel only.

ELIGIBILITY:
Inclusion Criteria:

* Physical findings suggestive of skin abscess warranting incision and drainage (determined by treating physician)

Exclusion Criteria:

* Abscess not suitable for drainage in the ED (eg. <1 cm induration, >15 cm induration)
* Immunocompromised status (eg. diabetic patient or taking immunosuppressive medication)
* Need for hospitalization following drainage
* Abscess located above the clavicles or significantly involving genitals/pilonidal region
* Previous instrumentation to the abscess
* Primary language not English or Spanish
* High probability of loss to follow up (parent does not commit to both mandatory follow up appointments)

Ages: 29 Days to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 81 (Actual)
Dates: Start 2014-09; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Treatment failure | 14 days
  Requiring reinstrumentation of abscess, or hospital admission for IV antibiotics

SECONDARY OUTCOMES:
Parental satisfaction with procedure | 1 Day
  Likert Scale of 1-5
Physician satisfaction with procedure | 1 Day
  Likert Scale of 1-5
Level of anxiety with wound care at home | 14 Days
  Likert Scale of 1-5
Level of simplicity with wound care at home | 14 Days
  Likert Scale of 1-5
Cosmetic success | 14 Days
  Hollander scale evaluating wound margins for step off, irregularity, wide separation, inversion
Parental satisfaction with scar | 90 Days
  Likert Scale of 1-5
Pain reduction with drainage procedure | 1 Day
  Revised FACES scale of 0-10
Frequency of post-drainage visits to a physician | 14 Days
  Any return for follow-up, packing removal, failure to improve, or any concern

CONTACTS AND LOCATIONS:
Overall Officials: Logan R Rencher, DO, Principal Investigator — UT-Austin Dell Children's Medical Center PEM Fellowship
Locations (1):
- Dell Children's Medical Center, Austin, Texas, United States

REFERENCES:
- [Background] Llera JL, Levy RC. Treatment of cutaneous abscess: a double-blind clinical study. Ann Emerg Med. 1985 Jan;14(1):15-9. doi: 10.1016/s0196-0644(85)80727-7. PMID 3880635
- [Background] Duong M, Markwell S, Peter J, Barenkamp S. Randomized, controlled trial of antibiotics in the management of community-acquired skin abscesses in the pediatric patient. Ann Emerg Med. 2010 May;55(5):401-7. doi: 10.1016/j.annemergmed.2009.03.014. Epub 2009 May 5. PMID 19409657
- [Background] Schmitz GR, Bruner D, Pitotti R, Olderog C, Livengood T, Williams J, Huebner K, Lightfoot J, Ritz B, Bates C, Schmitz M, Mete M, Deye G. Randomized controlled trial of trimethoprim-sulfamethoxazole for uncomplicated skin abscesses in patients at risk for community-associated methicillin-resistant Staphylococcus aureus infection. Ann Emerg Med. 2010 Sep;56(3):283-7. doi: 10.1016/j.annemergmed.2010.03.002. Epub 2010 Mar 26. PMID 20346539
- [Background] Leinwand M, Downing M, Slater D, Beck M, Burton K, Moyer D. Incision and drainage of subcutaneous abscesses without the use of packing. J Pediatr Surg. 2013 Sep;48(9):1962-5. doi: 10.1016/j.jpedsurg.2013.01.027. PMID 24074675
- [Background] Kessler DO, Krantz A, Mojica M. Randomized trial comparing wound packing to no wound packing following incision and drainage of superficial skin abscesses in the pediatric emergency department. Pediatr Emerg Care. 2012 Jun;28(6):514-7. doi: 10.1097/PEC.0b013e3182587b20. PMID 22653459
- [Background] O'Malley GF, Dominici P, Giraldo P, Aguilera E, Verma M, Lares C, Burger P, Williams E. Routine packing of simple cutaneous abscesses is painful and probably unnecessary. Acad Emerg Med. 2009 May;16(5):470-3. doi: 10.1111/j.1553-2712.2009.00409.x. Epub 2009 Apr 10. PMID 19388915
- [Background] Tsoraides SS, Pearl RH, Stanfill AB, Wallace LJ, Vegunta RK. Incision and loop drainage: a minimally invasive technique for subcutaneous abscess management in children. J Pediatr Surg. 2010 Mar;45(3):606-9. doi: 10.1016/j.jpedsurg.2009.06.013. PMID 20223328
- [Background] McNamara WF, Hartin CW Jr, Escobar MA, Yamout SZ, Lau ST, Lee YH. An alternative to open incision and drainage for community-acquired soft tissue abscesses in children. J Pediatr Surg. 2011 Mar;46(3):502-6. doi: 10.1016/j.jpedsurg.2010.08.019. PMID 21376200
- [Background] Ladd AP, Levy MS, Quilty J. Minimally invasive technique in treatment of complex, subcutaneous abscesses in children. J Pediatr Surg. 2010 Jul;45(7):1562-6. doi: 10.1016/j.jpedsurg.2010.03.025. PMID 20638546
- [Background] Alder AC, Thornton J, McHard K, Buckins L, Barber R, Skinner MA. A comparison of traditional incision and drainage versus catheter drainage of soft tissue abscesses in children. J Pediatr Surg. 2011 Oct;46(10):1942-7. doi: 10.1016/j.jpedsurg.2011.05.025. PMID 22008332
- [Background] Wright TN, Gilligan L, Zhurbich O, Davenport DL, Draus JM Jr. Minimally invasive drainage of subcutaneous abscesses reduces hospital cost and length of stay. South Med J. 2013 Dec;106(12):689-92. doi: 10.1097/SMJ.0000000000000032. PMID 24305529
- [Background] Hicks CL, von Baeyer CL, Spafford PA, van Korlaar I, Goodenough B. The Faces Pain Scale-Revised: toward a common metric in pediatric pain measurement. Pain. 2001 Aug;93(2):173-183. doi: 10.1016/S0304-3959(01)00314-1. PMID 11427329
- [Background] Tsze DS, von Baeyer CL, Bulloch B, Dayan PS. Validation of self-report pain scales in children. Pediatrics. 2013 Oct;132(4):e971-9. doi: 10.1542/peds.2013-1509. Epub 2013 Sep 2. PMID 23999954
- [Background] Singer AJ, Arora B, Dagum A, Valentine S, Hollander JE. Development and validation of a novel scar evaluation scale. Plast Reconstr Surg. 2007 Dec;120(7):1892-1897. doi: 10.1097/01.prs.0000287275.15511.10. PMID 18090752
- [Derived] Rencher L, Whitaker W, Schechter-Perkins E, Wilkinson M. Comparison of Minimally Invasive Loop Drainage and Standard Incision and Drainage of Cutaneous Abscesses in Children Presenting to a Pediatric Emergency Department: A Prospective, Randomized, Noninferiority Trial. Pediatr Emerg Care. 2021 Oct 1;37(10):e615-e620. doi: 10.1097/PEC.0000000000001732. PMID 30839438